CLINICAL TRIAL: NCT02531035
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Net Clinical Benefit of Sotagliflozin as Adjunct to Insulin Therapy in Type 1 Diabetes
Brief Title: A Phase 3 Study to Evaluate the Safety of Sotagliflozin in Patients With Type 1 Diabetes Who Have Inadequate Glycemic Control With Insulin Therapy Alone
Acronym: inTandem3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-312-T1DM; LX4211.312 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-08-20; First posted 2015-08-21 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus (T1DM); High Level of Sugar (Glucose) in the Blood
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Two placebo-matching to sotagliflozin tablets daily, orally, before the first meal of the day for 24 weeks.
  Interventions: Drug: Placebo
- Sotagliflozin 400 mg (Experimental): Sotagliflozin 400 milligram (mg) (two 200 mg tablets) once daily, orally, before the first meal of the day for 24 weeks.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin, once daily, before the first meal of the day
  Other Names: LX4211
  Arms: Sotagliflozin 400 mg
Drug: Placebo — Placebo, once daily, before the first meal of the day
  Arms: Placebo

SUMMARY:
This Phase 3 study was designed to demonstrate the net benefit of sotagliflozin versus placebo in patients with Type 1 Diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

* Participants had given written informed consent to participate in the study in accordance with local regulations
* Adult participants 18 years and older with a diagnosis of T1DM made at least 1 year prior to informed consent
* Participants were being treated with insulin or insulin analog
* Willing and able to perform self-monitoring of blood glucose (SMBG) and complete the study diary as required per protocol
* At the Screening Visit, A1C was between 7.0% to 11.0%
* Females of childbearing potential used an adequate method of contraception and had a negative pregnancy test

Exclusion Criteria:

* Use of antidiabetic agent other than insulin or insulin analog at the time of screening
* Use of sodium-glucose cotransporter (SGLT) inhibitors within 8 weeks prior to screening
* Chronic systemic corticosteroid use
* Type 2 diabetes mellitus (T2DM), or severely uncontrolled T1D as determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1405 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Sawhney, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (118):
- United States (33):
  - Lexicon Investigational Site, Concord, California
  - Lexicon Investigational Site, Escondido, California
  - Lexicon Investigational Site, La Jolla, California
  - Lexicon Investigational Site, San Marcos, California
  - Lexicon Investigational Site, Ventura, California
  - Lexicon Investigational Site, Walnut Creek, California
  - Lexicon Investigational Site, Aurora, Colorado
  - Lexicon Investigational Site, New Haven, Connecticut
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, West Palm Beach, Florida
  - Lexicon Investigational Site, Atlanta, Georgia
  - Lexicon Investigational Site, Macon, Georgia
  - Lexicon Investigational Site, Roswell, Georgia
  - Lexicon Investigational Site, New Orleans, Louisiana
  - Lexicon Investigational Site, Rockville, Maryland
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, Bloomfield Hills, Michigan
  - Lexicon Investigational Site, Omaha, Nebraska
  - Lexicon Investigational Site, Las Vegas, Nevada
  - Lexicon Investigational Site, Albany, New York
  - Lexicon Investigational Site, The Bronx, New York
  - Lexicon Investigational Site, Asheville, North Carolina
  - Lexicon Investigational Site, Chapel Hill, North Carolina
  - Lexicon Investigational Site, Greenville, North Carolina
  - Lexicon Investigational Site, Morehead City, North Carolina
  - Lexicon Investigational Site, Grand Forks, North Dakota
  - Lexicon Investigational Site, Bend, Oregon
  - Lexicon Investigational Site, Sioux Falls, South Dakota
  - Lexicon Investigational Site, Austin, Texas
  - Lexicon Investigational Site, San Antonio, Texas
  - Lexicon Investigational Site, Shavano Park, Texas
  - Lexicon Investigational Site, Salt Lake City, Utah
  - Lexicon Investigational Site, Seattle, Washington
- Argentina (2):
  - Lexicon Investigational Site, Córdoba, Córdoba Province
  - Lexicon Investigational Site, Buenos Aires
- Australia (9):
  - Lexicon Investigational Site, Coffs Harbour, New South Wales
  - Lexicon Investigational Site, Merewether, New South Wales
  - Lexicon Investigational Site, St Leonards, New South Wales
  - Lexicon Investigational Site, Wollongong, New South Wales
  - Lexicon Investigational Site, Herston, Queensland
  - Lexicon Investigational Site, Keswick, South Australia
  - Lexicon Investigational Site, Box Hill, Victoria
  - Lexicon Investigational Site, Fitzroy, Victoria
  - Lexicon Investigational Site, Parkville, Victoria
- Belgium (3):
  - Lexicon Investigational Site, Aalst
  - Lexicon Investigational Site, Ghent
  - Lexicon Investigational Site, Sint-Niklaas
- Bulgaria (5):
  - Lexicon Investigational Site, Plovdiv
  - Lexicon Investigational Site, Rousse
  - Lexicon Investigational Site, Smolyan
  - Lexicon Investigational Site, Sofia
  - Lexicon Investigational Site, Varna
- Canada (10):
  - Lexicon Investigational Site, Vancouver, British Columbia
  - Lexicon Investigational Site, Halifax, Nova Scotia
  - Lexicon Investigational Site, Barrie, Ontario
  - Lexicon Investigational Site, London, Ontario
  - Lexicon Investigational Site, Markham, Ontario
  - Lexicon Investigational Site, Oakville, Ontario
  - Lexicon Investigational Site, Thornhill, Ontario
  - Lexicon Investigational Site, Toronto, Ontario
  - Lexicon Investigational Site, Saint-Laurent, Quebec
  - Lexicon Investigational Site, Sherbrooke, Quebec
- Colombia (2):
  - Lexicon Investigational Site, Atlántico
  - Lexicon Investigational Site, Cundinamarca
- Czechia (4):
  - Lexicon Investigational Site, Krnov
  - Lexicon Investigational Site, Olomouc
  - Lexicon Investigational Site, Ostrava
  - Lexicon Investigational Site, Prague
- France (2):
  - Lexicon Investigational Site, Corbeil-Essonnes
  - Lexicon Investigational Site, Pierre-Bénite
- Germany (5):
  - Lexicon Investigational Site, Mainz, Palatinate
  - Lexicon Investigational Site, Sulzbach, Rosenberg Bavaria
  - Lexicon Investigational Site, Münster, Westphalia
  - Lexicon Investigational Site, Aschaffenburg
  - Lexicon Investigational Site, Aßlar
- Hungary (5):
  - Lexicon Investigational Site, Budapest
  - Lexicon Investigational Site, Eger
  - Lexicon Investigational Site, Esztergom
  - Lexicon Investigational Site, Győr
  - Lexicon Investigational Site, Sátoraljaújhely
- Israel (5):
  - Lexicon Investigational Site, Holon
  - Lexicon Investigational Site, Petach-Tikvah
  - Lexicon Investigational Site, Petah Tikva
  - Lexicon Investigational Site, Rehovot
  - Lexicon Investigational Site, Tel Litwinsky
- Italy (5):
  - Lexicon Investigational Site, Bologna
  - Lexicon Investigational Site, Catania
  - Lexicon Investigational Site, Latina
  - Lexicon Investigational Site, Milan
  - Lexicon Investigational Site, Rome
- New Zealand (7):
  - Lexicon Investigational Site, Epsom, Auckland
  - Lexicon Investigational Site, Takapuna, Auckland
  - Lexicon Investigational Site, Christchurch, Canterbury
  - Lexicon Investigational Site, Dunedin, Otago
  - Lexicon Investigational Site, Newtown, Wellington Region
  - Lexicon Investigational Site, Christchurch
  - Lexicon Investigational Site, Otahuhu
- Poland (4):
  - Lexicon Investigational Site, Gdynia
  - Lexicon Investigational Site, Katowice
  - Lexicon Investigational Site, Lublin
  - Lexicon Investigational Site, Warsaw
- Slovakia (3):
  - Lexicon Investigational Site, Bardejov
  - Lexicon Investigational Site, Bratislava
  - Lexicon Investigational Site, Levice
- South Africa (6):
  - Lexicon Investigational Site, Goodwood, Cape Town
  - Lexicon Investigational Site, Middelburg, Mpumalanga
  - Lexicon Investigational Site, Bloemfontein
  - Lexicon Investigational Site, Cape Town
  - Lexicon Investigational Site, Johannesburg
  - Lexicon Investigational Site, Port Elizabeth
- Spain (3):
  - Lexicon Investigational Site, Barcelona
  - Lexicon Investigational Site, Málaga
  - Lexicon Investigational Site, Seville
- United Kingdom (5):
  - Lexicon Investigational Site, Dundee, Scotland
  - Lexicon Investigational Site, Blackburn
  - Lexicon Investigational Site, Guildford
  - Lexicon Investigational Site, Leicester
  - Lexicon Investigational Site, Northampton

REFERENCES:
- [Derived] Garg SK, Henry RR, Banks P, Buse JB, Davies MJ, Fulcher GR, Pozzilli P, Gesty-Palmer D, Lapuerta P, Simo R, Danne T, McGuire DK, Kushner JA, Peters A, Strumph P. Effects of Sotagliflozin Added to Insulin in Patients with Type 1 Diabetes. N Engl J Med. 2017 Dec 14;377(24):2337-2348. doi: 10.1056/NEJMoa1708337. Epub 2017 Sep 13. PMID 28899222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 133 investigative sites across 19 countries: Poland, Slovakia, Spain, United Kingdom, Belgium, Bulgaria, Czech Republic, France, Germany, Hungary, Italy, Argentina, Australia, Canada, Colombia, Israel, New Zealand, South Africa and United States from 18 September 2015 to 18 April 2017.
Pre-assignment Details: 1405 participants with a diagnosis of Type 1 Diabetes were enrolled equally in 1 of 2 treatment groups: placebo or sotagliflozin 400 milligrams (mg).
Groups:
- Sotagliflozin 400 mg: Sotagliflozin 400 mg (two 200 mg tablets) once daily, orally, before the first meal of the day for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 400 mg
Started | 705 | 700
Treated | 703 | 699
Completed | 624 | 605
Not Completed | 81 | 95
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Noncompliance with study drug | 8 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 16 | 45
Not completed — Other | 3 | 2
Not completed — Withdrawal by Subject | 42 | 32
Not completed — Lost to Follow-up | 8 | 10
Not completed — Randomized, not treated | 2 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified Intent-to-treat (mITT) population included all randomly assigned participants who had taken at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 703 | 699 | 1402
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (14.04) | 43.3 (14.17) | 42.8 (14.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364 | 341 | 705
  Male | 339 | 358 | 697
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 5 | 7 | 12
  Black or African American | 22 | 24 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 621 | 619 | 1240
  Other | 37 | 31 | 68
  Not Applicable | 13 | 16 | 29
hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: percentage of A1C] — Population: A1C is the measurement of hemoglobin A1C. Data is available for 701 participants in the Placebo arm and 699 participants in the Sotagliflozin arm.
  percentage of A1C
    number analyzed (Participants) | 701 | 699 | 1400
    (all) | 8.21 (0.921) | 8.26 (0.965) | 8.23 (0.943)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 81.55 (17.032) | 82.40 (17.131) | 81.97 (17.081)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 19.6 (12.07) | 20.5 (12.37) | 20.0 (12.22)
Baseline Total Daily Insulin [Mean (Standard Deviation); unit: International units per kilogram (IU/kg)] | 0.71 (0.291) | 0.69 (0.276) | 0.70 (0.284)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2 (kilogram(s)/square meter)] | 28.10 (5.183) | 28.29 (5.128) | 28.19 (5.155)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With A1C <7.0% at Week 24 and No Episode of Severe Hypoglycemia and No Episode of Diabetic Ketoacidosis (DKA) After Randomization
Description: The primary composite endpoint included blood samples for the assessment of Hemoglobin A1C to determine the participants with a value <7.0%. A central blinded adjudication process determined whether participants experienced either DKA or Severe Hypoglycemia.
Time Frame: Week 24
Population: The primary efficacy analyses were based on the modified Intent-to-Treat (mITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 703 | 699
percentage of participants | 15.2 | 28.6
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values from Cochran-Mantel-Haenszel test stratified by different levels of stratification factors of BMI at Screening(<25 kg/m^2,>=25 kg/m^2),Week -2 A1C(<=9.0%, >9.0%),and using continuous subcutaneous insulin infusion(CSII) at Screening(yes,no); Percentage difference = 13.4, 95% CI 2-sided [8.97 to 17.81]

2. Secondary Outcome: Change From Baseline in A1C
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. Least Squares (LS) means were obtained from a mixed-effects model for repeated measures (MMRM) model including all available post baseline data. A negative change from Baseline (a lower AIC value at Week 24) indicates an improvement.
Time Frame: Baseline to Week 24
Population: Analyses included participants from the mITT population. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of A1c
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 628 | 627
percentage of A1c | -0.33 (0.031) | -0.79 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Testing according to hierarchical procedure. Post-Baseline LS means and p-values were obtained from MMRM model with treatment, randomization stratum of BMI at Screening (<25 kg/m^2, >=25 kg/m^2), randomization stratum of Week -2 A1C (<=9.0%, >9.0%), randomization stratum of use of CSII at Screening (yes, no), time (study week), and a treatment-by-time interaction as fixed categorical effects, and Baseline A1C-by-time interaction as a covariate; Test type: Superiority; p < 0.001, MMRM; Least Squares Mean Difference = -0.46, 95% CI 2-sided [-0.54 to -0.38]

3. Secondary Outcome: Absolute Change From Baseline in Body Weight
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model. A negative change from Baseline indicates a loss in body weight from Baseline to Week 24.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 633 | 630
kilograms (kg) | 0.77 (0.122) | -2.21 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Testing according to hierarchical procedure. Post-Baseline LS means and p-values were obtained from MMRM model with treatment, randomization stratum of BMI at Screening (<25 kg/m^2, >=25 kg/m^2), randomization stratum of Week -2 A1C (<=9%, >9%), randomization stratum of Use of CSII at Screening (Yes, No), time (study week), and a treatment-by-time interaction as fixed categorical effects, and Baseline weight-by-time interaction as a covariate; Test type: Superiority; p < 0.001, MMRM; Least squares mean difference = -2.98, 95% CI 2-sided [-3.31 to -2.66]

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) in the Subset of Participants With Baseline SBP >=130 Millimeter of Mercury (mmHg)
Description: An automatic sphygmomanometer was used with instructions on blood pressure measurements to allow for standardization. Week 16 was used because the protocol required Investigators to keep participant's hypertensive medications stable between Baseline and Week 16, unless a change was required for safety reasons. Baseline was defined as the last value collected prior to the first does of double-blind study medication. LS means were obtained from MMRM model including all available post baseline values. A negative change indicates a decrease in SBP between Baseline and Week 16.
Time Frame: Baseline to Week 16
Population: Participants from mITT population and who had a Baseline SBP >= 130 mm Hg. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 192 | 186
mmHg | -5.7 (0.90) | -9.2 (0.92)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Testing according to the hierarchical procedure. Post-Baseline LS means and p-values were obtained from MMRM model with treatment, randomization stratum of BMI at Screening (<25 kg/m2, >=25 kg/m2), randomization stratum of Week -2 A1C (<=9.0%, >9.0%), randomization stratum of use of CSII at Screening (yes, no), time (study week), and a treatment-by- time interaction as fixed categorical effects, and Baseline SBP-by-time interaction as a covariate; Test type: Superiority; p = 0.002, MMRM; Least Squares Mean Difference = -3.5, 95% CI 2-sided [-5.7 to -1.3]

5. Secondary Outcome: Percent Change From Baseline in Mean Daily Bolus Insulin Dose
Description: The mean bolus insulin dose in international units/day (IU/day) for Week 24 was the average over the 3 to 5 days prior to the Week 24 visit. The Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model including all available post Baseline values. A negative percent change from Baseline indicated a reduction in the amount of bolus insulin used and a positive percent change from Baseline indicated an increase in the amount of bolus insulin used between Baseline and Week 24.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change in IU/day
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 623 | 617
percent change in IU/day | 6.62 (2.272) | -5.71 (2.289)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Testing according to hierarchical procedure. Post-Baseline LS means and p-values were obtained from MMRM model with treatment, randomization stratum of BMI at Screening (<25 kg/m2, >=25 kg/m2), randomization stratum of Week -2 A1C (<=9.0%, >9.0%), randomization stratum of use of CSII at Screening (yes, no), time (study week), a treatment-by-time interaction as fixed categorical effects, and Baseline mean daily bolus insulin dose-by-time interaction as a covariate; Test type: Superiority; p < 0.001, MMRM; Least squares mean difference = -12.32, 95% CI 2-sided [-18.17 to -6.48]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to 30 days after end of treatment (Up to 28 Weeks)
Description: Analysis performed on safety population which includes participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 0/703 | 1/699
Serious Adverse Events (participants affected / at risk) | 23/703 | 48/699
Other Adverse Events (participants affected / at risk) | 70/703 | 70/699
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=703) | Sotagliflozin 400 mg (N=699)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Blood ketone body increased (Investigations) | 0 (0) | 1 (1)
Urine ketone body present (Investigations) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 4 (4) | 1 (1)
Encephalomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Aural polyp (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 (5) | 22 (26)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=703) | Sotagliflozin 400 mg (N=699)
Diarrhoea (Gastrointestinal disorders) | 17 (22) | 35 (41)
Viral upper respiratory tract infection (Infections and infestations) | 55 (62) | 41 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT02531035/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02531035/SAP_001.pdf